CLINICAL TRIAL: NCT03259490
Title: Bioequivalence of a Fixed Dose Combination Tablet of Empagliflozin/Linagliptin/Metformin Extended Release Compared to the Free Combination of Empagliflozin, Linagliptin, and Metformin Extended Release Tablets Following Oral Administration in Healthy Male and Female Subjects (an Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Study)
Brief Title: This Study Tests Whether Taking the Medicines Empagliflozin, Linagliptin, and Metformin Together in 1 Pill is the Same as Taking Them in Separate Pills. The Study is Done in Healthy Men and Women and Measures the Amount of Each Medicine in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1361-0003; 2017-000425-12 (EudraCT Number)
Record Dates: First submitted 2017-08-22; First posted 2017-08-23 (Actual); Results first posted 2020-02-21 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — empagliflozin; Linagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Treatment (Experimental): High dose empagliflozin/linagliptin/metformin XR fixed dose combination tablet
  Interventions: Drug: Empagliflozin/linagliptin/metformin HCl
- Reference Treatment (Experimental): Single tablets of empagliflozin + linagliptin + metformin XR
  Interventions: Drug: Empagliflozin; Drug: Linagliptin; Drug: Metformin HCl

INTERVENTIONS:
Drug: Empagliflozin/linagliptin/metformin HCl — Once daily
  Other Names: TRIJARDY® XR
  Arms: Test Treatment
Drug: Empagliflozin — Once daily
  Arms: Reference Treatment
Drug: Linagliptin — Once daily
  Arms: Reference Treatment
Drug: Metformin HCl — Once daily
  Arms: Reference Treatment

SUMMARY:
To establish the bioequivalence of one fixed dose combination (FDC) tablet of empagliflozin/linagliptin/metformin extended release (XR) versus the free combination of empagliflozin tablet, linagliptin tablet, and metformin XR tablets administered as a single dose under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Female subjects of childbearing potential willing to use adequate contraception.
* Further inclusion criteria apply

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR), or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (BPM)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to include healthy male and female subjects in this randomised, open label study. They were recruited from the volunteers' pool of the study site.
Pre-assignment Details: This trial was a two-way crossover study. All subjects received the 2 treatments in randomised order.
Groups:
- Test/ Reference (TR): Subjects were orally administered a single dose of 25 milligram (mg) empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 millilitre (mL) of water after a high-fat, high-calorie breakfast followed by a wash-out period of at least 35 days and then orally administered the free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast.
- Reference/ Test (RT): Subjects were orally administered the free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin extended release tablets with 240 mL of water after a high-fat, high-calorie breakfast followed by a wash-out period of at least 35 days and then orally administered a single dose of 25 milligram (mg) empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 millilitre (mL) of water after a high-fat, high-calorie breakfast.
Period: Period 1
Arm/Group | Test/ Reference (TR) | Reference/ Test (RT)
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2
Arm/Group | Test/ Reference (TR) | Reference/ Test (RT)
Started | 15 | 14
Completed | 14 | 14
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects who were documented to have received one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test/ Reference (TR) | Reference/ Test (RT) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: TS
  years | 37.1 (12.2) | 43.5 (8.0) | 40.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: TS
  Participants
    Female | 5 | 8 | 13
    Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not reported in this trial Population: TS
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 15 | 15 | 30
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz) for Empagliflozin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) for empagliflozin.
  Plasma concentrations and/or parameters of a subject were to be considered as non-evaluable,if for example:
  * The subject experienced emesis that occurred at or before 2 times median tmax of the respective treatment (median tmax was to be determined excluding the subjects experiencing emesis)
  * A predose concentration was >5% Cmax value of that subject
  * Missing samples/concentration data at important phases of pharmacokinetic (PK) disposition curve.
  Pharmacokinetic parameter set (PKS): This subject set included all subjects in the treated set (TS) who provided at least one primary or secondary PK parameter that was not excluded according to the description above. Thus, a subject was to be included in the PKS even if he/she contributed only one PK parameter value for one period to the statistical assessment.
Time Frame: Pharmacokinetic samples were collected at 1:30 hours: minutes pre dose and 0:30, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 5:00, 6:00, 7:00, 8:00, 10:00, 12:00, 24:00, 34:00, 48:00 and 72:00 hours:minutes post dose
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nanomoles*hours/ litres (nmol*h/L)
Groups:
- Empagliflozin/Linagliptin/Metformin FDC (Test): Subjects were orally administered a single dose of 25 mg empagliflozin/5 mg linagliptin/1000 mg metformin extended release (XR) fixed dose combination (FDC) tablet with 240 mL of water after a high-fat, high-calorie breakfast
- Empagliflozin/Linagliptin/Metformin FC (Reference): Subjects were orally administered a single dose of free combination of 25 mg empagliflozin, 5 mg linagliptin and 2 times 500 mg metformin XR tablets with 240 mL of water after a high-fat, high-calorie breakfast
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
nanomoles*hours/ litres (nmol*h/L) | 5656.07 (1.04) | 5488.31 (1.04)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); The assessment of bioequivalence was based upon two-sided 90% confidence intervals (CIs) for the ratios of the geometric means (test/reference) for the endpoints using an acceptance range of 80.00 to 125.00%; Test type: Other; ANOVA; Analysis of Variance (ANOVA) on the logarithmic scale including effects for 'sequence', 'subjects within sequences', 'period', and 'treatment'; Adjusted gmean ratio T/R (%) = 103.06, 95% CI 2-sided [100.36 to 105.83], Standard Deviation 5.8 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

2. Primary Outcome: AUC0-tz for Metformin.
Description: AUC0-tz for metformin.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nanogram*hours/ millilitres (ng*h/mL)
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
nanogram*hours/ millilitres (ng*h/mL) | 12455.82 (1.05) | 12412.57 (1.05)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gmean ratio T/R (%) = 100.35, 95% CI 2-sided [96.11 to 104.77], Standard Deviation 9.5 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

3. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to 72 Hours (AUC0-72) for Linagliptin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 hours (AUC0-72) for Linagliptin
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol*h/L
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
nmol*h/L | 238.84 (1.04) | 238.11 (1.04)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gmean ratio T/R (%) = 100.31, 95% CI 2-sided [96.65 to 104.10], Standard Deviation 8.2 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

4. Primary Outcome: Maximum Measured Concentration of the Empagliflozin in Plasma (Cmax)
Description: Maximum measured concentration of the empagliflozin in plasma (Cmax)
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol/L
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
nmol/L | 540.01 (1.04) | 540.26 (1.04)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gmean ratio T/R (%) = 99.95, 95% CI 2-sided [94.52 to 105.70], Standard Deviation 12.4 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

5. Primary Outcome: Cmax for Metformin in Plasma
Description: Cmax for metformin in plasma.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: ng/mL
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
ng/mL | 1237.16 (1.04) | 1147.88 (1.04)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gmean ratio T/R (%) = 107.78, 95% CI 2-sided [102.52 to 113.31], Standard Deviation 11.0 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

6. Primary Outcome: Cmax for Linagliptin in Plasma
Description: Cmax for linagliptin in plasma.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol/L
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
nmol/L | 5.69 (1.04) | 5.86 (1.04)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gmean ratio T/R (%) = 97.17, 95% CI 2-sided [92.63 to 101.93], Standard Deviation 10.6 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

7. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity) for Empagliflozin (AUC(0-∞)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) for Empagliflozin (AUC(0-∞)
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol*h/L
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
nmol*h/L | 5727.20 (1.04) | 5554.37 (1.04)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gmean ratio T/R (%) = 103.11, 95% CI 2-sided [100.38 to 105.92], Standard Deviation 5.9 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

8. Secondary Outcome: AUC(0-∞) for Metformin
Description: AUC(0-∞) for Metformin
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: ng*h/mL
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
ng*h/mL | 12745.62 (1.05) | 12724.27 (1.05)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gmean ratio T/R (%) = 100.17, 95% CI 2-sided [95.68 to 104.86], Standard Deviation 10.1 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

9. Secondary Outcome: AUC(0-∞) for Linagliptin
Description: AUC(0-∞) for Linagliptin
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Standard Error); unit: nmol*h/L
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
Number analyzed (Participants) | 29 | 29
nmol*h/L | 384.27 (1.05) | 394.95 (1.05)
Statistical Analysis 1: Comparison: Empagliflozin/Linagliptin/Metformin FDC (Test) vs Empagliflozin/Linagliptin/Metformin FC (Reference); [analysis description as in outcome 1, analysis 1]; Test type: Other; ANOVA; [statistical method as in outcome 1, analysis 1]; Adjusted gmean ratio T/R (%) = 97.30, 95% CI 2-sided [91.65 to 103.29], Standard Deviation 13.2 — The standard deviation is actually intra-individual geometric co-efficient of variation (gCV)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) which occurred through the treatment phase and throughout the residual effect period (REP); up to 50 days
Description: REP for the combined treatment with empagliflozin, linagliptin, and metformin, when measurable drug levels or pharmacodynamic effects were still likely to be present, was defined as 7 days after the last administration of trial medication.
Arm/Group | Empagliflozin/Linagliptin/Metformin FDC (Test) | Empagliflozin/Linagliptin/Metformin FC (Reference)
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 11/29 | 6/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin/Linagliptin/Metformin FDC (Test) (N=29) | Empagliflozin/Linagliptin/Metformin FC (Reference) (N=29)
Nausea (Gastrointestinal disorders) | 1 | 2
Oral herpes (Infections and infestations) | 2 | 0
Headache (Nervous system disorders) | 8 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT03259490/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03259490/SAP_001.pdf